CLINICAL TRIAL: NCT03528174
Title: Assessment of a Novel Sensing Catheter During Automated Insulin Delivery in Patients With Type 1 Diabetes
Brief Title: Single Hormone Closed Loop Study With PDT Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Castle, Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18241
Record Dates: First submitted 2018-04-26; First posted 2018-05-17 (Actual); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Hormone closed loop (Experimental): Subjects will have glucose managed using the Artificial Pancreas Control system (APC) using insulin only. Insulin will be infused through the Pacific Diabetes Technologies CGM Insulin Infusion system.
  Interventions: Device: Artificial Pancreas Control system (APC); Device: Pacific Diabetes Technologies CGM Insulin Infusion system

INTERVENTIONS:
Device: Artificial Pancreas Control system (APC) — This intervention is a single hormone closed loop system including a Nexus 5 smart phone, two tslim insulin pumps, a Dexcom G5 CGM and two PDT glucose sensing cannulas that together make up a new experimental, investigational device system. The algorithm included in the APC is an automated version of the Fading Memory Proportional Derivative (FMPD) insulin and glucagon control algorithm.
Device: Pacific Diabetes Technologies CGM Insulin Infusion system — An integrated combination CGM/insulin infusion system

SUMMARY:
The study described within this protocol is designed to test a single hormone closed-loop algorithm for managing blood glucose in type 1 diabetes using insulin only and a new device for measuring glucose continuously in the immediate vicinity of subcutaneous insulin delivery. Subjects will undergo one all day closed loop study using insulin only. The closed loop insulin only system includes a Dexcom G5 transmitter, a Nexus 5 smart phone and two Tandem tslim pumps connected to two Pacific Diabetes Technologies glucose sensing cannulas. The closed loop system will be started after G5 2 hour sensor start-up with an IV catheter for frequent blood withdrawal for 10 hours.

DETAILED DESCRIPTION:
Subjects will undergo one 12 hour inpatient study. During this intervention visit, subjects will wear the single hormone closed loop system which includes two t:slim insulin pumps to deliver insulin or saline through two investigational PDT glucose sensing cannulas, and a Dexcom G5 CGM to measure glucose. The subject will come to the research center at approximately 7am for the inpatient visit. The Dexcom G5 sensor and PDT glucose sensing cannulas will be placed after arrival. An 18-22 gauge IV catheter will be placed for blood sampling every 15 minutes after sensor warm-up is complete for measuring blood glucose concentration. After a 2 hour warm-up period for the G5 sensor, glucose will be controlled using the FMPD single hormone mode. The single hormone mode of the controller determines insulin delivery rates based on proportional and derivative error through one t:slim insulin pump. The second t:slim insulin pump will deliver normal saline at the same delivery rates as the insulin. Subjects will eat breakfast and lunch at approximately 11 am and 3 pm respectively. Subjects will have the ability to complete light exercise on a treadmill. The closed loop system will be stopped at approximately 6pm with removal of all devices.

During the study, the subject will wear one subcutaneous DexcomTM G5 continuous glucose monitoring (CGM) system. The CGM system will provide sensed glucose data every 5 minutes. The accuracy of the sensed data will be obtained by reference measurements of two YSI venous blood glucose values to calibrate the sensor at the beginning of the closed loop study. Sensed glucose data will be wirelessly transmitted via Bluetooth Low Energy (BTLE) from the Dexcom G5 transmitter to the Nexus 5 master controller every five minutes. The controller is a Google Nexus 5 phone. The smart phone will wirelessly communicate via BTLE to two Tandem t:slim insulin pumps, one for automated insulin delivery and one of automated saline delivery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 21 to 65 years of age.
* Current use of an insulin pump for at least 3 months with stable insulin pump settings for > 2 weeks.
* HbA1c ≤ 10% at screening.
* Body Mass Index ≥ 22.
* Total daily insulin requirement is less than 200 units/day.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as reported by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* Hematocrit of less than 36% for men, less than 32% for women.
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator.
* History of Diabetic Ketoacidosis during the prior 6 months prior to screening visit, as diagnosed on hospital admission or as judged by the investigator.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to lispro insulin.
* Allergy to acrylate-based skin adhesives.
* Need for uninterrupted treatment of acetaminophen.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Beta blockers or non-dihydropyridine calcium channel blockers.
* Current use of any medication intended to lower glucose other than insulin (ex. use of liraglutide).
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the subject's safety or compliance with the protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Castle, MD, Principal Investigator — Oregon Health and Science University; Peter Jacobs, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Hormone Closed Loop
Started | 10
Completed | 8
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — sensors dislodged | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Relative Difference of Sensed Glucose Values
Description: Assess the mean absolute relative difference for the PDT CGM/insulin infusion system based on all reference YSI venous blood glucose values.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: percentage of reference blood glucose
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
percentage of reference blood glucose | 13.5 (4.6)

2. Secondary Outcome: Percent of Time With Sensed Glucose Between 70-180 mg/dl
Description: Assess the percent of time with sensed glucose between 70-180 mg/dl based on the Dexcom G5 CGM sensor values for all subjects.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
percentage of time | 59.8 (27.42)

3. Secondary Outcome: Percent of Time With Sensed Glucose Less Than 70 mg/dl
Description: Assess the percent of time with sensed glucose less than 70 mg/dl based on the Dexcom G5 CGM sensor values for all subjects.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
percentage of time | 3.3 (7)

4. Secondary Outcome: Percent of Time With Sensed Glucose Less Than 54 mg/dl
Description: Assess the percent of time with sensed glucose less than 54 mg/dl based on the Dexcom G5 CGM sensor values for all subjects.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
percentage of time | 0.3 (0.7)

5. Secondary Outcome: Percent of Time With Sensed Glucose Greater Than 250 mg/dl
Description: Assess the percent of time with sensed glucose greater than 250 mg/dl based on the Dexcom G5 CGM sensor values for all subjects.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
percentage of time | 12.4 (17.7)

6. Secondary Outcome: Mean Sensed Glucose
Description: Assess the average sensor glucose based on the Dexcom G5 CGM sensor values.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
mg/dL | 167.8 (71)

7. Secondary Outcome: Number of Carbohydrate Treatments
Description: Assess the average number of carbohydrate treatments per study defined as 15 or 20 grams of carbohydrates.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: carbohydrate treatments
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
carbohydrate treatments | 0.6 (1.9)

8. Secondary Outcome: Mean Amount of Insulin Delivered
Description: Assess the average amount of insulin delivered per study in units/kg.
Time Frame: up to 10 hours
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
units/kg | 0.24 (0.11)

9. Secondary Outcome: Mean Score of Visual Analog Scale at 15 Minutes
Description: Assess the average score on the visual analog scale at 15 minutes after insertion of the PDT glucose sensor. This scale will be used to measure sensor site discomfort from the PDT glucose sensing cannula. The subject completes the visual analog scale by drawing a single vertical line through a 100 mm line corresponding to the perceived intensity (severity) of discomfort from the insertion of the sensors. Subjects will be instructed to mark their line starting on the left side over to the right side. If subjects are feeling no discomfort, they would circle the vertical line on the left end of the scale. If subjects are currently feeling the worst discomfort possible, they would circle the vertical line on the right side of the scale. One staff member will measure all scales and document score as a measurement of 0-100.
Time Frame: 15 minutes post insertion
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
mm | 6.4 (8.3)

10. Secondary Outcome: Mean Score of Visual Analog Scale at 120 Minutes
Description: Assess the average score on the visual analog scale at 120 minutes after insertion of the PDT glucose sensor.This scale will be used to measure sensor site discomfort from the PDT glucose sensing cannula. The subject completes the visual analog scale by drawing a single vertical line through a 100 mm line corresponding to the perceived intensity (severity) of discomfort since the devices were inserted. Subjects will be instructed to mark their line starting on the left side to the right side. If subjects are feeling no discomfort, they would circle the vertical line on the left end of the scale. If subjects are currently feeling the worst discomfort possible, they would circle the vertical line on the right side of the scale. One staff member will measure all scales and document score as a measurement of 0-100.
Time Frame: 120 minutes post insertion
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
mm | 0.7 (1.3)

11. Secondary Outcome: Mean Score of Visual Analog Scale at End of Study
Description: Assess the average score on the visual analog scale at the end of the study. This scale will be used to measure sensor site discomfort from the PDT glucose sensing cannula. The subject completes the visual analog scale by drawing a single vertical line through a 100 mm line corresponding to the perceived intensity (severity) of discomfort since the devices were inserted. Subjects will be instructed to mark their line starting on the left side to the right side. If subjects are feeling no discomfort, they would circle the vertical line on the left end of the scale. If subjects are currently feeling the worst discomfort possible, they would circle the vertical line on the right side of the scale. One staff member will measure all scales and document score as a measurement of 0-100.
Time Frame: End of 10 hour study
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
mm | 8.9 (21.7)

12. Secondary Outcome: Mean Draize Scale for Erythema for the Left Sensing Cannula at End of Study for All Subjects
Description: Assess the average score on the Draize scale at the end of the study of the PDT glucose sensor. The investigator discharging the subject will inspect each PDT glucose sensing cannula insertion site and rate the level of redness (erythema) and swelling (edema). Both the left and right insertion sites will be inspected. Erythema will be measured from 0-4. A score of 0 indicates no erythema, a score of 1 indicates very slight, barely perceptible erythema, a score of 2 indicates well defined erythema, a score of 3 indicates moderate erythema, and a score of 4 indicates severe erythema, beet redness to slight eschar formation. Edema will be measured from a score of 0-4. A score of 0 indicates no edema, a score of 1 indicates very slight, barely perceptible edema, a score of 2 indicates well defined edema, a score of 3 indicates moderate edema, raised approximately 1 mm, and a score of 4 indicates severe edema, raised greater than 1 mm and beyond exposure area.
Time Frame: End of 10 hour study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
units on a scale | 0.2 (0.4)

13. Secondary Outcome: Mean Draize Scale for Edema for the Left Sensing Cannula at End of Study for All Subjects
Description: as for outcome 12
Time Frame: end of 10 hour study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
units on a scale | 0.15 (0.37)

14. Secondary Outcome: Mean Draize Scale for Erythema for the Right Sensing Cannula at End of Study for All Subjects
Description: as for outcome 12
Time Frame: End of 10 hour study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
units on a scale | 0.2 (0.4)

15. Secondary Outcome: Mean Draize Scale for Edema for the Left Sensing Cannula at End of Study for All Subjects
Description: as for outcome 12
Time Frame: end of 10 hour study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Hormone Closed Loop
Number analyzed (Participants) | 10
units on a scale | 0.2 (0.4)

ADVERSE EVENTS:
Time Frame: Up to 10 hours
Arm/Group | Single Hormone Closed Loop
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Hormone Closed Loop (N=10)
hospitalization for emesis (Gastrointestinal disorders) | 1 (1) — Hospitalization for persistant emesis and nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03528174/Prot_SAP_000.pdf